CLINICAL TRIAL: NCT05883423
Title: Application of Frailty Prevention Care Management Program on Frailty and Health Function of Community Elderly Adults
Brief Title: Application of Frailty Prevention Care Management Program of Community Elderly Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin Chia Hui, PHD,RN,Associate Professor, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202202269B0
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Frailty
Keywords: elderly adults; frailty prevention care management programs
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPCMP-Old Age group (Experimental): The program mainly refers to Ha and Park (2020), and extends the development of the 12-week FPCMP-Old Age program, which combines sports and health integrated nursing management courses (nutrition, psychosocial, drug and other health management activities). Twice a week, 2 hours each time, 12 weeks, a total of 24 times, the execution period is scheduled to be from July to the end of September.
  Interventions: Other: FPCMP-Old Age
- usual group (No Intervention): Participate in the original health promotion activities of the community group

INTERVENTIONS:
Other: FPCMP-Old Age — 1. Exercise program：The main purpose of the exercise program is to improve cardiorespiratory endurance, upper and lower limb muscle strength and endurance, body flexibility, sense of balance and coordination. The exercise program is carried out with a suspension training system, which can improve core muscle strength, improve physical fitness, activate more core and stabilizing muscle groups, increase joint stability, and strengthen ligaments.
  2. Health integrated nursing management courses (nutrition, psychosocial, drug and other health management activities involved)
  Arms: FPCMP-Old Age group

SUMMARY:
This study first explored the relationship between basic demographic variables, frailty and health function of community-based adults and elderly. Promote and explore the effect of the Frailty Prevention Care Management Program (FPCMP-Old Age) on the frailty and health function of the elderly in the community.

The elderly in the long-term care community bases in the central and southern regions were selected as the object of acceptance. The study design is divided into two years(Two phases) study, the first phase is to develop a 12-week frailty prevention care management plan (FPCMP-Old Age). The second stage is to introduce FPCMP-Old Age to carry out a pilot study in the south-central community. A total of 70 cases were accepted in the experimental group and the control group. This study was divided into two groups, which were grouped by convenient sampling. The experimental group underwent the FPCMP-Old Ag program; the control group only maintained the original site to delay disability and dementia activities. In this study, pre-intervention, post-intervention, and four-week follow-up were conducted, and three questionnaires were evaluated. Each time it was estimated to spend 30 minutes for each answer, the activity lasted for 12 weeks. The execution period this time is from January 1, 2023 to December 30, 2024, but the time for accepting cases is from June 1, 2023 to December 31, 2023. There are four research tools in this study, namely: demographic variables, chronic disease and health problem scale, frailty detection tool (TFI-T), health function (refer to the 2016 recommendation of the Ministry of Education and Sports Administration for the fitness of the elderly group Test items, testing the subject's body composition, upper and lower limb muscle strength, upper and lower limb flexibility, cardiorespiratory endurance, dynamic and static balance) and nutritional status (mini nutritional assessment) and other tools. Data were collected in triplicate, and generalized estimating equations were used to analyze whether there were differences in interaction effects between groups, within groups, and time.

The Frailty Prevention Care Management Program (FPCMP-Old Age) can help community-based adults and older adults reduce frailty and improve health function.

DETAILED DESCRIPTION:
Background ：The elderly are a high-risk group for developing frailty symptoms. The prevalence of frailty ranges from 16% for those over 65 years of age to 52% for those over 85 years of age, and it increases proportionally with age. Frailty is not a disease. It represents the cumulative functional degeneration of various systems. It is a sub-healthy state or a stage before disability. Some elderly people have different degrees of frailty. In mild cases, there may be no clinical symptoms. Interference part of life; more severe cases may lead to disability or disease.

Objective：This study first explored the relationship between basic demographic variables, frailty and health function of community-based adults and elderly. Promote and explore the effect of the Frailty Prevention Care Management Program (FPCMP-Old Age) on the frailty and health function of the elderly in the community.

Methods：The elderly in the long-term care community bases in the central and southern regions were selected as the object of acceptance. The study design is divided into two years(Two phases) study, the first phase is to develop a 12-week frailty prevention care management plan (FPCMP-Old Age). The second stage is to introduce FPCMP-Old Age to carry out a pilot study in the south-central community. A total of 70 cases were accepted in the experimental group and the control group. This study was divided into two groups, which were grouped by convenient sampling. The experimental group underwent the FPCMP-Old Ag program; the control group only maintained the original site to delay disability and dementia activities. In this study, pre-intervention, post-intervention, and four-week follow-up were conducted, and three questionnaires were evaluated. Each time it was estimated to spend 30 minutes for each answer, the activity lasted for 12 weeks. The execution period this time is from January 1, 2023 to December 30, 2024, but the time for accepting cases is from June 1, 2023 to December 31, 2023. There are four research tools in this study, namely: demographic variables, chronic disease and health problem scale, frailty detection tool (TFI-T), health function (refer to the 2016 recommendation of the Ministry of Education and Sports Administration for the fitness of the elderly group Test items, testing the subject's body composition, upper and lower limb muscle strength, upper and lower limb flexibility, cardiorespiratory endurance, dynamic and static balance) and nutritional status (mini nutritional assessment) and other tools. Data were collected in triplicate, and generalized estimating equations were used to analyze whether there were differences in interaction effects between groups, within groups, and time.

Conclusions/practical application： The Frailty Prevention Care Management Program (FPCMP-Old Age) can help community-based adults and older adults reduce frailty and improve health function.

ELIGIBILITY:
Inclusion Criteria:

* Community elders over 60 years old; able to communicate in Mandarin and Taiwanese and voluntarily participate in this course

Exclusion Criteria:

* Those who suffer from severe chronic diseases (such as heart disease, end-stage kidney disease, cancer) or severe illness, etc., and are unable to exercise
* Those who have severe visual and hearing impairments or use assistive devices without communication barriers
* Suffering from severe bone and joint diseases (for example: severe osteoporosis, severe knee or shoulder joint degeneration)
* Arrhythmia that requires drug treatment or a cardiac pacemaker
* Those with severe cognitive impairment.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The Taiwanese version of Tilburg frailty indicator(TFI-T) | It takes 5 minutes to fill out the questionnaire
  This scale was translated by the researchers and other teams from The Taiwanese version of Tilburg frailty indicator (TFI-T) developed by Gobbens and other scholars in 2010. It is divided into three parts, with a total of 15 items. The first part measures physical frailty (score range 0 -8 points), including: Unexpected weight loss, physical fitness, difficulty walking, balance, visual problems, hearing problems, hand strength, and physical fatigue. The second part is mental frailty (score range 0-4 points), including: cognition, depressive symptoms, anxiety and coping ability. The third part is social-level frailty (score range 0-3 points), including: living alone, social relationship and social support, etc., with 0-1 points for each question, and a total score of 15 points.
Chronic Disease and Health Problems Scale | It takes 5 minutes to fill out the questionnaire
  The research tools refer to the "Severity of Chronic Diseases and Health Problems" edited by Pan Baoxia (2012). There are 21 chronic diseases and health problems scales in total. Respondents are asked to self-evaluate their chronic diseases and The number of symptoms of health problems, and explore the severity of chronic diseases and health problems that interfere with daily life. The scoring method for the severity of interference is 0 points for "no inconvenience", 1 point for "slight inconvenience", and 2 points for "slight inconvenience". The total score ranges from 0 to 42 points. Chronic diseases or health problems affect life more seriously.
Health Function | It takes 15 minutes to test health function
  Refer to the Senior Fitness Test (SFT) recommended by the Sports Administration of the Ministry of Education in 2016, which refers to the ability of subjects to perform daily activities independently without excessive fatigue and safety concerns. The muscles of the elderly are tested separately. Strength, Muscular Endurance, Cardiorespiratory Endurance, Body Flexibility, Balance, Coordination, Reaction Time and Body Composition
Nutritional Assessment | It takes 5 minutes to fill out the questionnaire
  The Mini Nutritional Assessment-Short Form (MNA-SF) is used for assessment. MNA-SF has 6 questions, the minimum score range is 0-2 points, the maximum score range is 0-3 points, and the total score 14 points, if the score ≥ 11 points, it means that the nutritional status of the subject is within the acceptable range, 8-11 points: there is a risk of malnutrition, 0-7 points: malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hui Lin, PhD, Study Director — Chang Gung Medical Foundation
Locations (1):
- Taiwan, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulmez I. Effects of Angle Variations in Suspension Push-up Exercise. J Strength Cond Res. 2017 Apr;31(4):1017-1023. doi: 10.1519/JSC.0000000000001401. PMID 26950344
- [Result] Ha J, Park YH. Effects of a Person-Centered Nursing Intervention for Frailty among Prefrail Community-Dwelling Older Adults. Int J Environ Res Public Health. 2020 Sep 13;17(18):6660. doi: 10.3390/ijerph17186660. PMID 32933119
- [Result] McDermott AY, Mernitz H. Exercise and older patients: prescribing guidelines. Am Fam Physician. 2006 Aug 1;74(3):437-44. PMID 16913163